CLINICAL TRIAL: NCT02599428
Title: Recovery After ICU Treatment: A Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Stine Estrup, Junior Doctor, PhD Student, Zealand University Hospital
Other Study IDs: SE 1-16
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Delirium; Critical Illness; Quality of Life
MeSH Terms: conditions — Delirium; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This project aims to investigate the physical, mental and cognitive recovery after admission to the Intensive Care Unit (ICU).

This will be done by a three and 12 month follow up after discharge. The patients will be scored with four validated methods for evaluating their health related quality of life, anxiety and depression, cognitive function and physical impairments

DETAILED DESCRIPTION:
An increasing number of patients are treated at ICUs worldwide. The majority of these patients survive critical illness and are discharged from the hospital. A stay at the ICU is most often related to life-threatening conditions and displays a major impact on both physical and mental resources of the patients. Studies have shown that a great part of these patients also have physical and psychological impairments lasting for a long period after their hospital stay. The condition is termed the "post intensive care syndrome" (PICS) and describes a state with wide range of symptoms as fatigue, depression, anxiety, memory loss as well as both cognitive and physical impairment. During the first five years after discharge, more than half of ICU survivors had suffered at least one episode of depression or anxiety

ICU treatment often involves immobilization and sedation that may lead to both muscle weakness, critical illness myopathy and/or polyneuropathy. This may not only affect the patients during the ICU or hospital stay, but also for a longer post-discharge period. A recent study demonstrated that measured physical health related quality of life was impaired for up to one year after hospitalization, and that the physical performance at five years post-discharge continued to be lower than in the background population. The physical impairments may also influence patient's working ability, and among previously working individuals only half had returned to work within the first year after ICU hospitalization. After five years, up to 25 % still had not returned to work.

In Denmark, more than 30.000 people are annually admitted to intensive care units. The annual report from the Danish Intensive Care Database (DID) present data regarding a variety of outcomes, including length of stay, survival rate and 90 days re-admission to hospital. The reports demonstrate an increased quality of care but offer limited information on longer term outcome including quality of life for these patients. A recent study have indicated that Danish patients might suffer from the same psychological and physical impairments as found in international studies, but a better characteristic of the population is needed. Especially since the level of public care, including early rehabilitation in hospital differs between countries.

It is therefore essential to investigate and describe the needs, standard of care and the physical and cognitive status of these patients both in-hospital and post-discharge in order to establish the right level of aftercare for the Danish population. This study aims at investigating the in-hospital care as well as the physical and cognitive status of a Danish cohort of ICU patients at 3 and 12 month post-discharge.

The investigators plan to do a substudy regarding exposure to circadian light and delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Admitted to the ICU for > 24 h

Exclusion Criteria:

* Not able to speak and understand Danish
* Discharged from the ICU to terminal care
* Patients transferred to another hospital during ICU stay
* Patients living outside the Region of Zealand
* Patient with severe dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU at Zealand University Hospital, Køge, in the study period
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2016-02; Primary Completion 2018-03 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Cognitive function measured by Repeatable Battery for the Assessments of Neuropsychological Status (RBANS) | 3 months after discharge
  The Repeatable Battery for the Assessments of Neuropsychological Status (RBANS) evaluation status at 3 and 12 months after discharge from ICU

SECONDARY OUTCOMES:
Adherence to checklist based on rehabilitation guidelines | At discharge from hospital and 3 months
  Adherence to a checklist at discharge from ICU and hospital that evaluates rehabilitation efforts based on guidelines from NICE (the National Institute for Health and Care Excellence)
Health related quality of life measured by Short form health survey (SF 36) | 3 and 12 months
  Short form health survey (SF 36) score at 3 and 12 month follow up
Anxiety and depression measured by Hospital anxiety and depression scale (HADS) | 3 and 12 months
  Hospital anxiety and depression scale (HADS) score at 3 and 12 month follow up
Physical function measured by Chelsea critical care physical assessment tool (CPAx) | 3 and 12 months
  Chelsea critical care physical assessment tool (CPAx) at 3 and 12 month follow up
Mortality | At discharge from hospital (variable time) and at 90 days postdischarge
  All cause mortality
Delirium at the ICU measured by CAM-ICU | At discharge from ICU (variable time)
  Delirium during ICU stay, measured as days with a positive CAM-ICU score or CAM-ICU negative delirium treated with anti-psychotics
Consumption of opioids at admission and on follow up | At admission to hospital, at 3 month follow up
  Percentage of patients with a daily consumption of opioids (strong/weak) at hospital admission and at 90 days discharge
Consumption of anti-depressants before and after ICU stay | At admission to hospital, at 3 month follow up
  Percentage of patients with a daily consumption of anti-depressants at hospital admission and at 90 days after discharge
Receiving statins before and after ICU stay | At admission to hospital, at 3 month follow up
  Percentage of patients with a daily consumption of statins at hospital admission and at 90 days after discharge
Cognitive function measured by Repeatable Battery for the Assessments of Neuropsychological Status (RBANS) | 12 months after discharge
  The Repeatable Battery for the Assessments of Neuropsychological Status (RBANS) evaluation status at 3 and 12 months after discharge from ICU

CONTACTS AND LOCATIONS:
Overall Officials: Ole Mathiesen, MD, Study Chair — Zealand University Hospital, Køge Hospital
Locations (1):
- University Hospital Zealand, Køge, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Wolters A, Bouw M, Vogelaar J, Tjan D, van Zanten A, van der Steen M. The postintensive care syndrome of survivors of critical illness and their families. J Clin Nurs. 2015 Mar;24(5-6):876-9. doi: 10.1111/jocn.12678. Epub 2014 Dec 1. No abstract available. PMID 25441007
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Derived] Estrup S, Kjer CKW, Vilhelmsen F, Poulsen LM, Gogenur I, Mathiesen O. Physical function and actigraphy in intensive care survivors-A prospective 3-month follow-up cohort study. Acta Anaesthesiol Scand. 2019 May;63(5):647-652. doi: 10.1111/aas.13317. Epub 2019 Jan 8. PMID 30623414